CLINICAL TRIAL: NCT00822484
Title: Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ILV-095 Administered Subcutaneously to Healthy Japanese Male Subjects
Brief Title: Study Evaluating Single Doses of ILV-095 in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 3226K2-1001
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ILV-095 (Active Comparator): 6 SC single dose injections
  Interventions: Biological: ILV-095
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ILV-095
  Arms: ILV-095
Other: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of single doses of ILV-095 in healthy Japanese male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 20 to 45 years inclusive at screening. Sexually active men must agree to use a medically acceptable form of contraception during the study and continue it for 12 weeks after study drug administration.
* Body mass index (BMI) in the range of 17.6 to 26.4 kg/m2 and body weight greater than or equal to 45 kg.
* Healthy as determined by the investigator on the basis of screening evaluations.
* Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.
* Have a high probability for compliance with and completion of the study.

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Any subject who had orthopedic surgery within 12 weeks of the screening visit or has planned (elective) orthopedic surgery within 12 weeks of study drug administration.
* Acute disease state (eg, nausea, vomiting, infection, fever, active infection, or diarrhea) within 7 days before enrollment.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-02; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability will be evaluated from the reported AEs including any injection-site reactions, physical examinations, vital sign measurements, cardiac rhythm monitoring, 12-lead ECGs, and clinical laboratory test results. | 3 weeks per group

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 3 weeks per group

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3226K2-1001&StudyName=Study%20Evaluating%20Single%20Doses%20of%20ILV-095%20in%20Healthy%20Japanese%20Male%20Subjects